CLINICAL TRIAL: NCT03735654
Title: Assessing the Impact of Muscle Strength and Fatigability on Gait Performance Using Single Joint and Multi-joint Assessments in People With Multiple Sclerosis
Brief Title: Multi-joint Muscle Fatigability and Gait Performance in People With Multiple Sclerosis
Acronym: MS_Gait
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Harris-Love, Director, 3MAP Lab, and Assoc. Director, CRC Human Performance Research Unit, Washington D.C. Veterans Affairs Medical Center
Other Study IDs: 01931
Record Dates: First submitted 2018-10-03; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare walking to leg strength and endurance in people with multiple sclerosis (PwMS). Using these findings, we hope to be better understand what causes PwMS to have problems walking.

DETAILED DESCRIPTION:
The purposes of the research are to determine the association of gait performance with lower extremity muscle fatigability and strength measures, and create a preliminary model that can better explain the variance in gait performance based on these muscle performance values. Objective criterion-based measures of physical fatigue (i.e., fatigability) and muscle weakness have been associated with impaired task performance in people with multiple sclerosis (MS). MS-related deficits in muscle capacity result in higher fall risks and a loss of function. However, it is unclear if lower extremity fatigability tests add clinical value to objective strength testing in the rehabilitation and clinical management of MS. Better understanding how patterns of lower extremity (LE) fatigability and strength affect mobility in people with MS could improve outcome measure development and inform rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* History of multiple sclerosis
* Expanded Disability Status Scale < 7.0
* Receives care at the Washington DC Veteran's Affairs Medical Center Neurology Service and Multiple Sclerosis Center of Excellence - East

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive care at the Washington DC Veteran's Affairs Medical Center Neurology Service and Multiple Sclerosis Center of Excellence - East
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Performance (FAP) | 1 Day
  The FAP is used to quantify self-selected gait.
Hip, knee, and ankle fatigability | 1 Day
  For isometric tests, a exhaustion time will be calculated by determining the time that peak impulse declines to 50% using a method validated for individual with MS.
Hip, knee, and ankle maximal volitional contraction | 1 Day
  Maximal volitional contraction will be measured by the load cell using isometric expressed as peak torque.

SECONDARY OUTCOMES:
Adult Myopathy Assessment Tool (AMAT) | 1 Day
  The Adult Myopathy Assessment Tool (0-45 score) is a physical test battery used to evaluate functional performance in individuals with neuromuscular disease. The test consists of 13 measures for functional mobility, balance, strength and endurance to mimic activities of daily living.
5 times sit to stand test (5STS) | 1 Day
  The 5STS reflects the amount of time required for a participant to complete 5 sit to stand maneuvers without using their hands. For this study we used the 5STS as a measure of functional capacity in people with multiple sclerosis.

OTHER OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | 1 Day
  The MFIS is based on items derived from interviews with MS patients concerning how fatigue impacts their lives. This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The MFIS consists of 21 items and is a subscale of the MS Quality of Life Inventory.
Fatigue Severity Score (FSS) | 1 Day
  The FSS is a questionnaire that can indicate severe fatigue related to MS. Scores range from 9-63 with higher scores indicating higher levels of fatigue.
Neurology Quality of Life Adult Fatigue Bank (AFB) | 1 Day
  The AFB measures are a collection of patient- reported questionnaires and short forms developed with the goal of assessing health-related quality of life (HRQL) across all neurological disorders.
Activity Balance Confidence Score (ABC) | 1 Day
  The ABC Scale is a 16-item questionnaire that serves as a rating of self-perceived confidence during performance of activities of daily living. Scores range from 0-100 with higher scores indicating greater confidence.
BioSensic measure of Reciprocal Compensatory Index (RCI) | 1 Day
  BalanSens is a biosensor and is based on widely-available kinematic sensors (i.e. accelerometer, gyroscope and magnetometer). The system measures ankle and hip motion in three dimensions. It allows for object measurement of balance when a patient performs Romberg, sharpened Romberg eyes open and closed and single leg stance.
Multiple Sclerosis Spasticity Scale (MSSS-88) | 1 Day
  The MSSS-88 is a subjective assessment of day-to-day spasticity symptoms and functional impact in eight clinically separate areas. Scores range from 88-352 and higher scores indicate greater spasticity.
Kurtzke Expanded Disability Status Scale (EDSS) | 1 Day
  This is a standardized neurological disability scale developed specifically for MS. It accounts broadly for MS symptoms, including things like mobility, mental health, and sensory disturbances. Scores range from 0-10 with higher scores indicating loss of ambulatory ability.
Beck Depression Index II (BDI-II) | 1 Day
  The BDI-II is a widely used test for measuring depression among individuals.
Epworth Sleepiness Scale (ESS) | 1 Day
  The ESS is a subjective questionnaire that measures sleep disturbances and excessive sleepiness. Scores range from 0-24, with higher scores indicating greater daytime sleepiness.
Montreal Cognitive Assessment (MoCA) | 1 Day
  The MoCA is a subject questionnaire that can be used as a screening tool for cognitive dysfunction in people with MS.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc, Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States